CLINICAL TRIAL: NCT03276585
Title: Epidemiological Study on Insomnia and Depression Using Home Sleep Monitors in a Japanese Rural City Population
Brief Title: Night in Japan Home Sleep Monitoring Study
Acronym: NinJaSleep
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Shiga University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Koka city (Unknown)
Responsible Party: Sponsor
Other Study IDs: 29-111; UMIN000028675 (Registry Identifier: UMIN Clinical Trials Registry (UMIN-CTR), Japan)
Record Dates: First submitted 2017-09-03; First posted 2017-09-08 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Sleep Initiation and Maintenance Disorders; Depression
Keywords: home sleep monitor; Sleep Apnea Syndromes; questionnaire
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators hypothesized that depression is associated with home sleep EEG, subjective sleepiness and insomnia symptoms. To test this, the investigators plan to perform sleep examination with single channel EEG, in combination with questionnaire survey for insomnia, sleepiness, depression and job stress to Koka city government employees.

DETAILED DESCRIPTION:
Depression is a major global public health problem and is projected to carry an even greater burden of disease worldwide in the coming decades. Both insomnia and excessive daytime sleepiness (EDS) are sleep disturbance that commonly occur as a principal component of depression. However, studies analyzing objective measurements of EDS or insomnia were very limited. Multiple sleep latency test (MSLT, four nap studies under polytrophic recordings in sleep labs) in psychiatric diseases demonstrated highly heterogeneous results. This may come from most studies had small sample size, which is frequently associated with both depressive symptoms and sleepiness.

Full polysomnography (full-PSG) provides comprehensive information about sleep duration and architecture, but it is too expensive and too cumbersome for large-scale or repeated-measures evaluations (¥96,380/case by Diagnosis Procedure Combination/Per-Diem Payment System in Japan). Using in-laboratory full-PSG as the gold standard has limitations in validity, partly because participants tend to sleep more poorly in the laboratory than at home. Thus, full-PSG may be unsuitable for screening large populations or for repeated evaluations. Actigraphy is a simple method for monitoring locomotor activity and can be used to estimate sleep/wake time but cannot access sleep architecture and sleep staging. Recent advances in electronic technologies and sensor interfaces have enabled small sleep portable monitors. The investigators compared a newly developed single-channel EEG monitoring system (SleepWell Co. Ltd., Osaka, Japan) with simultaneously recorded polysomnography. Single-channel EEG showed reasonable agreement with full-PSG (percent agreement and kappa coefficient of sleep stages were 86.9% ± 4.42 and 0.75 ± 0.081, respectively). This single channel EEG may be suitable to monitor daily sleep more easily in epidemiological settings.

Objective sleep monitoring is important. In measuring excessive daytime sleepiness, for example, subjective evaluation (Epworth sleepiness scale) failed to show much correlation with objective measurements with polygraph recordings. Individuals at high risk for depression have been found to have negative biases in processing information. They may answer subjective insomnia measurements more severely. Previous studies on depression and insomnia came mainly from subjective measures, which may be influenced by such negative evaluation bias. Objective sleep EEG measurements may be useful in overcoming such biases.

Sleep epidemiological study is limited in Japan. For example, sound estimates of prevalence of sleep apnea syndrome in Japan were lacking: previous Japanese studies have been limited by use of nonprobability samples, low response rates, small samples, and other methodologic problems. The investigators have performed sleep epidemiological study in a male working population in Japan. In the study, sleep apnea syndrome (apnea-hypopnea index (AHI) or respiratory event index (REI) ≥15) in males was estimated as 22.3%, which was similar to those in other studies including Sleep Heart Health Study. However, its target population included only Japanese "males". Studies in Japanese females are still missing.

In Japan, employers have to perform annual medical check-ups to their employees including detailed blood biochemical examination. Adding sleep survey to such annual examination, the investigators can analyze detailed physical effects of sleep with minimal costs. Even after the survey, with these annual examinations, the investigators can analyze incidences of lifestyle-related diseases (hypertension, diabetes, dyslipidemia, etc.) in the future.

Recent studies suggest that Rapid eye movement (REM) sleep is important in emotional memory consolidation. REM sleep may be the key between emotional distress and mental disorders: such as insomnia, depression, and posttraumatic stress disorder. To elucidate these interactions, it is essential to perform epidemiological study with sleep EEG monitoring. Without EEG, the investigators cannot analyze REM sleep at all.

In this study, the investigators plan to analyze around 1,000 participants and analyze sleep EEG at home. This will make a big difference, because participants usually sleep poorer in sleep laboratory than at home.

The investigators have performed questionnaire surveys on insomnia and depression among local government employees in Koka, Shiga prefecture, Japan since 2014. The investigators have good relationship with Koka city government and participation rate to the surveys were as high as 93%, whose mean age was 42.0±10.3 years (range: 18-61 years) .

The investigators hypothesized that depression is associated with home sleep EEG, subjective sleepiness and insomnia symptoms. To test this, the investigators plan to perform sleep examination with single channel EEG, in combination with questionnaire survey for insomnia, sleepiness, depression and job stress to Koka city government employees.

The database, constructed during this project, will serve as fundamentals in the future studies in analyzing mental stress, insomnia, depression, lifestyle-related diseases and social costs in the general population. In the follow-up studies in the future, the investigators will also analyze cardio-vascular attach events, cerebrovascular attach events, sick leaves, incidents of depression and/or insomnia in the subgroups.

The investigators plan to get funding from Japanese ministry of education science and culture to perform home sleep apnea testing. Because sleep apnea is a very prevalent sleep disorder (over 20% of males have moderate-to-severe sleep apnea with 15 times per hour or more of apnea/hypopnea events). Participants usually wake up for a short period (arousal) after each apnea/hypopnea event, which cause sleep fragmentation in PSG/EEG. Sleep apnea syndrome is a risk factor for depressive symptoms and sleepiness.

When some part of this population (for example, 50% of participants with depression and similar number of those without) undergo clinical diagnostic interviews by psychiatrists, the investigators can use this data to develop diagnostic tool for depression in the future.

ELIGIBILITY:
Inclusion Criteria:

* Koka city government employees (Koka city, Shiga prefecture, Japan)

Exclusion Criteria:

* Subjects who need legally acceptable representative to consent.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Koka city government employees (Koka city, Shiga prefecture, Japan)
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-09-06 (Actual); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | 2 weeks
  The ISI is a seven-item self-rating scale. The subjects rate the severity of insomnia, the distress, and the functional impairment associated with insomnia.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | 2 weeks
  PHQ-9 is a 9-item self-administrated questionnaire, which assess Major depressive disorder.
Epworth Sleepiness Scale (ESS) | 2 weeks
  ESS is a 8-item self-administrated questionnaire, which assess the sleepiness.

OTHER OUTCOMES:
Single-channel Electroencephalogram (EEG) | 1 week
  Single-channel Electroencephalogram (EEG) can be used to analyze sleep latency, sleep efficiency and delta wave power at home. Sleep latency is the amount of time it takes to fall asleep after the lights have been turned off. Sleep efficiency is ratio of total sleep time to time in bed. EEG delta wave power is used as an index of the hypothetical sleep 'pressure' that has accumulated during wakefulness.
Respiratory Event Index (REI) | 1 week
  REI (numbers of apneas and hypopneas divided by recorded hours with home sleep testings), is used for diagnosis and severity definition of sleep apnea syndrome.
Chalder fatigue scale | 2 weeks
  Chalder fatigue scale is a self-rating score, which is now widely used to measure the severity of 'tiredness'.
General Anxiety Disorder-7 (GAD-7) | 2 weeks
  GAD-7 is a 7-item self-administrated questionnaire, which assess generalized anxiety disorder.
FIRST (Ford Insomnia Response to Stress Test) | 2 weeks
  FIRST is a 9-item self-rating score measuring the likelihood of the occurrence of sleep disturbances in response to commonly experienced stressful situations.
8-Item Short-Form Health Survey (SF-8) | 1 month
  The SF-8 is an 8-item self-administrated questionnaire, which assess health-related quality of life.
WHO Health and Work Performance Questionnaire (WHO-HPQ) | 1 month
  WHO-HPQ is a self-report instrument designed to estimate the workplace costs of health problems in terms of self-reported sickness absence (absenteeism) and reduced job performance (presenteeism).
The Brief Job Stress Questionnaire | 1 month
  The Brief Job Stress Questionnaire is a 57-item self-administrated questionnaire, which assess stress in workplace. Japanese government launched the Stress Check Program in 2015. The program recommends to use the Brief Job Stress Questionnaire for defining "high-stress" workers.
Athens Insomnia Scale (AIS) | 1 month
  AIS is an 8-item self-administrated questionnaire, which assess Insomnia.
the Circadian Energy Scale (CIRENS) | 2 weeks
  CIRENS is a very short and simple chronotype measurement tool based on energy.
Four-Variable Screening Tool | 2 weeks
  With knowledge of only 4 easily ascertainable variables, moderate-to-severe sleep apnea syndrome can be easily detected in clinical and public health settings (SLEEP 2009;32(7):939-948).

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Kadotani, MD,PhD, Principal Investigator — Department of Sleep and Behavioral Sciences, Shiga University of Medical Science
Locations (1):
- Shiga University of Medical Science, Ōtsu, Shiga, Japan

IPD SHARING:
Plan to Share IPD: Undecided
We have not decided with whom to collaborate.

REFERENCES:
- [Derived] Omichi C, Kaminishi Y, Kadotani H, Sumi Y, Ubara A, Nishikawa K, Matsuda A, Ozeki Y. Limited social support is associated with depression, anxiety, and insomnia in a Japanese working population. Front Public Health. 2022 Nov 21;10:981592. doi: 10.3389/fpubh.2022.981592. eCollection 2022. PMID 36483246